CLINICAL TRIAL: NCT05677828
Title: Effect of the Addition of Letrozole in in Vitro Fertilization (IVF) Following a Prior Failed IVF Cycle With an Antagonist or Short Protocol Without Letrozole
Brief Title: SMART Protocol vs Antagonist Protocol in IVF
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: CCER 21-22 - 21
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Diminished Ovarian Reserve
Keywords: IVF; Fertility issues
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antagonist - SMART: Women who have had a SMART IVF stimulation cycle with Letrozole after a failed antagonist IVF stimulation cycle between 2010 and 2020.
- Antagonist - Antagonist: Women who have had an antagonist stimulation IVF cycle after a previously failed antagonist IVF stimulation cycle between 2010 and 2020.

SUMMARY:
This retrospective study aims to assess the effect of adding letrozole in patients who have previously undergone an IVF cycle with either an antagonist or short protocol, with patients who have undergone a second cycle of IVF with an antagonist or short protocol without the addition of letrozole.

DETAILED DESCRIPTION:
A limited number of studies suggest that the addition of letrozole to gonadotropins for IVF is associated with an increase in oocyte count, blastocyst count and implantation rate. These differences are presumed to be caused by an increase in intra-ovarian androgens associated with the addition of letrozole.

In patients with reduced ovarian reserve or reduced oocyte quality in the previous cycle, supplementation with of letrozole has the potential to increase oocyte count or oocyte quality, thereby resulting in more transferable blastocysts. The antagonist stimulation protocol with the addition of letrozole is commonly referred to as the SMART protocol (Stimulation with Minimal Adverse effects, Retrieval and Transfer

ELIGIBILITY:
Inclusion Criteria for the SMART IVF protocol:

* Women between the ages of 20 and 42 inclusively
* Women proceeding with a SMART IVF protocol following an antagonist IVF protocol between 2010 and 2020 (study group) or women proceeding with an antagonist protocol following an antagonist IVF protocol between 2010 and 2020 (control group)
* Delay of 1 year between both IVF cycle

Exclusion Criteria:

* Women undergoing fertility preservation
* Oocyte donation IVF cycles
* Diagnosed severe male factor requiring surgical sperm extraction (micro-tese or TESA)

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: This retrospective cohort study will analyze IVF cycles in antagonist and SMART stimulation protocols during the period from 2010 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of utilizable blastocysts obtained | approximately 20 days
  Comparing 2 different IVF cycle protocols in terms of total dose of gonadotropins used

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hemmings, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada